CLINICAL TRIAL: NCT02262702
Title: Panadol Osteo PBS Claims Cohort Study
Brief Title: Panadol Osteo Pharmaceuticals Benefit Scheme (PBS) Claims Cohort Study
Status: Withdrawn | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 202175; RH01690 (Other: GSK)
Record Dates: First submitted 2013-05-23; First posted 2014-10-13 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Extended Release Paracetamol: Participants prescribed with extended release paracetamol tablet containing 665 mg paracetamol.
  Interventions: Drug: Paracetamol 665 mg
- Standard Paracetamol: Participants prescribed with standard paracetamol tablet containing 500 mg paracetamol.
  Interventions: Drug: Paracetamol 500 mg

INTERVENTIONS:
Drug: Paracetamol 665 mg — Paracetamol 665 mg tablet
  Other Names: Panadol Osteo
  Groups: Extended Release Paracetamol
Drug: Paracetamol 500 mg — Paracetamol 500 mg tablet
  Groups: Standard Paracetamol

SUMMARY:
The aim of this observational study is to compare the use of an extended release paracetamol formulation with standard paracetamol in a cohort of Australian concessional patients with osteoarthritis (OA), to assess differences in prescribing patterns and patient compliance.

DETAILED DESCRIPTION:
This retrospective analysis of physician prescribing data (long-term concessional cohort from the Medicare Australia PBS claims dataset for the time period 2008-2011 (4 years) will compare the use of extended release paracetamol (Panadol Osteo) with standard paracetamol 500mg in a cohort of Australian concessional patients with OA, to assess differences in prescribing patterns and patient compliance.

ELIGIBILITY:
Inclusion Criteria:

* Participants prescribed with a paracetamol product and categorized as a concessional patient
* Participants with new episodes of OA (no history of OA paracetamol in previous 12 months) or suffering from chronic OA (history of OA paracetamol in the previous 12 months)

Exclusion Criteria:

* Participants with Rheumatoid arthritis or other auto-immune inflammatory conditions
* Participants receiving the following anti-rheumatoid therapies:Immunimodulators such as methotrexate, leflunamide and TNF blockers
* Participants receiving treatment for cancer pain

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of Australian concessional patients with osteoarthritis
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Relative number of prescriptions of an extended release paracetamol formulation and a standard release paracetamol formulation. | January 2009 to December 2010
  Number of episodes of treatment for OA with the extended release formulation and the standard release formulatins will be counted.
Relative treatment compliance with an extended release paracetamol formulation and a standard release paracetamol formulation | January 2009 to December 2010
  Interval between the repeat doses of extended release paracetamol formulation and the standard release paracetamol formulation.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline